CLINICAL TRIAL: NCT02012855
Title: Effect of Exercise and Glycemic Index of Carbohydrate Feeding on Postprandial Lipid Metabolism
Brief Title: Effect of Different Types of Carbohydrates Consumed After Exercise on Blood Fat Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Collaborators: Heart and Stroke Foundation of Canada (Other)
Responsible Party: Principal Investigator, Phil Chilibeck, Ph.D., University of Saskatchewan
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 000041
Record Dates: First submitted 2013-08-15; First posted 2013-12-16 (Estimated); Last update posted 2017-05-05 (Actual); Status verified 2017-05

CONDITIONS: Hyperlipidemia
MeSH Terms: conditions — Hyperlipidemias | interventions — Exercise; Diet

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Exercise only (Experimental): 90 minutes of exercise
  Interventions: Behavioral: Exercise
- Exercise and high glycemic index meal (Experimental): 90 minutes of exercise followed by a high glycemic index meal matched for calories expended during the exercise
  Interventions: Behavioral: Exercise; Other: Diet (meal type)
- Exercise and low glycemic index meal (Experimental): 90 minutes of exercise followed by a low glycemic index meal matched for calories expended during the exercise
  Interventions: Behavioral: Exercise; Other: Diet (meal type)
- No exercise and no meal (No Intervention): No exercise and no meal

INTERVENTIONS:
Behavioral: Exercise
  Arms: Exercise and high glycemic index meal; Exercise and low glycemic index meal; Exercise only
Other: Diet (meal type)
  Arms: Exercise and high glycemic index meal; Exercise and low glycemic index meal

SUMMARY:
The increase in fat (i.e. triglyceride) in the blood after a meal is a well-established risk factor for heart disease (Nordestgaard et al. 2007). Endurance exercise is beneficial for improving the blood lipid response to a subsequent meal; that is, the appearance of fat (triglyceride) in the blood is less after a meal if endurance exercise was performed shortly before (i.e. within half a day) of the meal (Petit et al. 2003). This benefit of exercise is unfortunately negated if the after-exercise food choice to replace the calories expended during exercise is one containing high glycemic index carbohydrates. For example, if a high glycemic index carbohydrate is consumed after an evening exercise session, the exercise no longer has an effect of lowering triglyceride in the blood after a meal consumed the next morning (Harrison et al. 2009; Burton et al. 2008). Very rarely do people perform an exercise session and then fast until their next meal hours later. The more common practice is to consume food immediately after the exercise to enhance recovery and because hunger is stimulated with exercise. Consuming carbohydrate with a low glycemic index has been shown to reduce the level of fat in the blood following a subsequent meal (Gruendel et al. 2007). To date, no studies have examined the effects of consuming a low-glycemic index meal after exercise on the blood fat response to a subsequent meal. The specific objective of our research is to determine the effect of consuming low glycemic index lentils after an endurance exercise session on the blood fat (triglyceride) response to a subsequent meal. Twenty-five overweight or obese men will have their blood triglycerides measured four times over six hours after a high-fat morning meal following four different conditions, in a randomized, counterbalanced, cross-over design (i.e. the 25 subjects will each participate in all four conditions, where the order of conditions for each person is randomized): 1) After exercise (90 minutes of moderate intensity walking) is performed the evening before, followed by caloric replacement with a high-glycemic index meal (i.e. white bread and instant mashed potatoes); 2) After the same exercise is performed the evening before, followed by caloric replacement with a lentil-based meal; 3) After the same exercise is performed the evening before, followed by fasting; 4) After a no exercise/ no meal condition (i.e. control condition). In addition to measuring blood triglycerides we will measure blood insulin, free fatty acid, high density lipoproteins, low density lipoproteins, and glucose levels as these are also related to cardiovascular disease risk and may be altered with exercise and lentil consumption. We will also measure the muscle's ability to burn fat (i.e. fat oxidation) by assessing respiratory gases (oxygen consumption and carbon dioxide output) after the high-fat meal because we expect exercise and lentils to increase fat oxidation. Our expected results are that consuming lentils after endurance exercise will lower the blood triglyceride response to a subsequent meal compared to exercise alone or when high-glycemic index carbohydrates are consumed after the exercise.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index of 25 or greater
* 18-44 years of age

Exclusion Criteria:

* diabetics
* smokers
* those taking medications for cholesterol or glucose

Ages: 18 Years to 44 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2013-08; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Change in blood triglycerides | Change from baseline at 6 hours

SECONDARY OUTCOMES:
Change in blood glucose | Change from baseline at 6 hours
Change in fat oxidation | Change from baseline at 6 hours
Change in low density lipoproteins | Change from baseline at 6 hours
Change in high density lipoproteins | Change from baseline at 6 hours
Change in total cholesterol | Change from baseline at 6 hours
Change in insulin level | Change from baseline at 6 hours

CONTACTS AND LOCATIONS:
Overall Officials: Philip D Chilibeck, Ph.D., Principal Investigator — University of Saskatchewan
Locations (1):
- University of Saskatchewan, Saskatoon, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No